CLINICAL TRIAL: NCT01959191
Title: Clinical Significance of Platelet Reactivity on Clopidogrel During Off-pump Coronary Artery Bypass
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0309
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
Keywords: Platelet activity, CABG, off-pump surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low platelet reactivity group: Platelet reactivity will be measured after 7-days treatment of clopidogrel by VerifyNow system and the cohort will be divided by two group according to P2Y12 reactivity unit (PRU) cutoff value. Receiver operating characteristic (ROC) curves will be plotted to assess the optimal PRU cutoff value for differentiating between patients with and without subsequent MACEs after 1 year of follow-up. Low platelet reactivity indicates good response to clopidogrel and high platelet reactivity, resistance to clopidogrel. Groups will be "Low platelet reactivity group" and "High platelet reactivity group"
  Interventions: Drug: Dual antiplatelet therapy including aspirin and clopidogrel after off-pump coronary bypass surgery
- high platelet reactivity group: Platelet reactivity will be measured after 7-days treatment of clopidogrel by VerifyNow system and the cohort will be divided by two group according to P2Y12 reactivity unit (PRU) cutoff value. Receiver operating characteristic (ROC) curves will be plotted to assess the optimal PRU cutoff value for differentiating between patients with and without subsequent MACEs after 1 year of follow-up. Low platelet reactivity indicates good response to clopidogrel and high platelet reactivity, resistance to clopidogrel. Groups will be "Low platelet reactivity group" and "High platelet reactivity group"
  Interventions: Drug: Dual antiplatelet therapy including aspirin and clopidogrel after off-pump coronary bypass surgery

INTERVENTIONS:
Drug: Dual antiplatelet therapy including aspirin and clopidogrel after off-pump coronary bypass surgery — aspirin 100mg/day and clopidogrel 75mg/day, PO, from the day of surgery for 1 year

SUMMARY:
Objective: To evaluate the early and late prognoses of patients according to platelet reactivity after clopidogrel administration and determine whether the measurement of platelet inhibition predicted 1-year clinical outcomes after off-pump coronary bypass (OPCAB) Study design

* Prospective, observational, single-center study
* Subjects with OPCAB surgery who meet all inclusion and exclusion criteria will be enrolled.
* Platelet reactivity after 7-days clopidogrel treatment from the day of surgery will be measured by VerifyNow system.
* Dual antiplatelet therapy including aspirin and clopidogrel will be administered for 1 year after surgery and subjects will be followed-up for 1 year about primary endpoint.
* Cutoff value of P2Y12 reactivity units (PRUs) for primary endpoint will be assessed and the cohort will be divided by the PRU cutoff value (low/high platelet reactivity groups).
* The primary and secondary endpoints will be compared between two groups

ELIGIBILITY:
Inclusion Criteria:

* Patients with indications for surgical myocardial revascularization
* Patients who undergo off-pump coronary artery bypass
* Age between 19~80 years
* Patients with signed informed consent

Exclusion Criteria:

* Patients with combined surgery with coronary bypass grafting
* On-pump conversion
* Patients with moderate renal dysfunction (creatinine>2.0mg/dl) or need for dialysis
* Patients with chronic treatment with proton pump inhibitors
* Patients with preoperative bleeding
* Thrombocytopenia (Platelet count 70,000/ml)
* Re-do surgery
* Early death before the measurement of platelet reactivity

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with indications for surgical myocardial revascularization
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2008-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACEs) | 1 year after off-pump coronary bypass surgery
  The primary endpoint of the study was the 1-year incidence of MACEs, which included the following: (1) cardiac death, defined as death in the presence of acute coronary syndrome, sudden cardiac arrest with documented cardiac arrhythmia, or refractory congestive heart failure; 2) nonfatal MI; and (3) target vessel revascularization in relation to platelet reactivity as measured by the VerifyNow system.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiovascular Surgery, Severance Cardiovascular Hospital , Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Patti G, Nusca A, Mangiacapra F, Gatto L, D'Ambrosio A, Di Sciascio G. Point-of-care measurement of clopidogrel responsiveness predicts clinical outcome in patients undergoing percutaneous coronary intervention results of the ARMYDA-PRO (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty-Platelet Reactivity Predicts Outcome) study. J Am Coll Cardiol. 2008 Sep 30;52(14):1128-33. doi: 10.1016/j.jacc.2008.06.038. PMID 18804738